CLINICAL TRIAL: NCT03396471
Title: Single-arm Phase 2 Study to Examine Pembrolizumab and Concurrent Radiation to Induce an Abscopal Effect in Patients With Previously Treated Carcinoma of Unknown Primary (CUP16-268)
Brief Title: Study of Pembrolizumab and Concurrent Radiation in Patients With Previously Treated Carcinoma of Unknown Primary
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study failed to meet its interim analysis endpoint
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN CUP16-268
Record Dates: First submitted 2017-12-27; First posted 2018-01-11 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Unspecified Site
MeSH Terms: conditions — Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Assignment (Experimental): Pembrolizumab + External Beam Radiation Therapy
  Interventions: Drug: Pembrolizumab; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV at day -21, then day 1 of each 21-day cycle for a maximum of 24 continuous months of Pembrolizumab (35 cycles) from Cycle 1 Day 1 (C1D1) can be administered.
  Other Names: Keytruda
Radiation: External Beam Radiation Therapy — 20-30 Gy over five fractions for up to two cycles.
  Other Names: External Beam Radiation Therapy (EBRT)

SUMMARY:
Single-arm phase 2 study to examine pembrolizumab and concurrent radiation to induce an abscopal effect in patients with previously treated carcinoma of unknown primary (CUP16-268)

DETAILED DESCRIPTION:
This is a proof-of-principle single-arm phase 2 study in patients with previously treated CUP. All patients receive pembrolizumab combined with Radiation Therapy (RT) to a metastatic site, so as to induce an abscopal tumor response. The treatment combination will be repeated with RT delivery to a second metastatic site in a non-overlapping RT field.

The results will be compared with historical control. The primary endpoint is the confirmed response rate (RR) in a non-irradiated site based on best responding abscopal lesion. This study will also evaluate the following secondary endpoints: RR in a non-irradiated site based on RECIST 1.1, adverse events, progression-free survival (PFS), overall survival (OS), time-to-progression (TTP), and disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 within 28 days prior to registration.
* Archival tissue must be available and identified during screening and shipped prior to Day -21. If archival tissue is not available and the subject is not undergoing a standard of care biopsy, the subject must undergo a research biopsy to obtain fresh tissue prior to start of treatment.
* Carcinoma of unknown primary after the following diagnostic procedures have been performed if clinically indicated and are unrevealing of the primary site:

  * Complete history and clinically appropriate physical
  * CT scan of chest, abdomen, and pelvis
  * Directed evaluation of symptomatic areas
  * Mammogram in women
  * Colonoscopy in patients with liver metastasis or an elevated CEA
  * Direct pathologic comparison with prior tumor specimens, where possible, even if prior tumor is early-stage or clinically remote from current disease NOTE: Immunohistochemical stains will be performed according to institutional standards. If a primary carcinoma is identified, the patient should undergo treatment as appropriate for that primary tumor and not be enrolled in the study. The above diagnostic workup does not need to be performed if: (1) it was previously completed at the time of original diagnosis or (2) the investigator does not believe the workup has clinical utility at the current time, given that the patient has received interval therapy.
* Histologic confirmation of metastatic adenocarcinoma, poorly differentiated non-small cell carcinoma, or poorly differentiated squamous carcinoma. NOTE: Pathology consultation at Mayo Clinic is recommended if clinically indicated. One scenario is where unknown primary is the most likely diagnosis but immunostains show relatively site-specific marker staining (e.g., CD45, TTF1, chromogranin, GATA3, PAX8, PSA, melanocytic markers). Information provided for pathology consultation should include recent H&P and imaging reports.
* If and when available, submission of genomic sequencing and expression profiling results is mandatory. Results of testing are not required prior to treatment.
* At least one measurable lesion (per RECIST 1.1) outside the planned RT fields.
* Stable or progressive disease after, or was unable to tolerate, at least one line of prior anticancer therapy for this disease. NOTE: For patients with stable disease, it is strongly encouraged to confirm the presence of active disease (eg, demonstrating 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) avidity via PET or repeat biopsy).
* Radiation oncology consultation at enrolling site ≤ 56 days prior to registration to confirm at least two metastatic lesions which are targetable by RT at doses and schedule prescribed in this study and which reside in non-overlapping RT fields.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration.

  * Hematological

    * Absolute Neutrophil Count (ANC) ≥ 900 K/mm3
    * Hemoglobin (Hgb) ≥ 8.5 g/dL without transfusion or EPO dependency (≤ 7 days prior to assessment)
    * Platelets ≥ 90,000 / mcL
  * Renal

    ---Creatinine OR Calculated creatinine clearance: ≤ 1.5 X upper limit of normal (ULN) OR

    ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Hepatic

    * Bilirubin Total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN OR total bilirubin ≤2 X ULN if liver metastases are present
    * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
    * Albumin > 2.5 g/dL
* Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to registration. NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: breast milk cannot be stored for future use while the mother is being treated on study
* Females of childbearing potential and males must be willing to abstain from heterosexual activity (abstinence) or use effective methods of contraception as described in the protocol from the time of informed consent until 120 days after treatment discontinuation. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Willingness to return to the enrolling institution for follow up
* Willingness to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Prior radiation to an area of the body which, if included in the current radiation field, poses an unacceptably high risk of toxicity in the opinion of the investigator. NOTE: A prior field that overlaps with the current field, by itself, does not exclude the patient.
* Any of the following

  --Melanoma. NOTE: Positive tumor staining for S-100 or HMB45 alone does not exclude patients.

  ---If immunostains are performed, and any of the below tests are positive:
  * Hematologic CD45+ (others such as CD2, CD20, CD30, CD43 also suggest hematologic origin)
  * Lung or thyroid origin (Thyroid Transcription Factor [TTF-1]). NOTE: Patients with biopsy proven TTF-1 positive tumor who do not have clinical evidence for either lung or thyroid cancer (e.g. a dominant lung mass) are still eligible.
* Progressed on 4 or more lines of prior chemotherapy for this cancer. NOTE: Bisphosphonates and neoadjuvant/adjuvant anticancer therapies (including locally directed therapies) do not count as a line of therapy with regard to this exclusion criteria.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. NOTE: Inhaled steroids or steroid injections for joint disease are allowed.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Prior severe allergic reactions to a monoclonal antibody or hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Other active malignancy which requires current treatment and which in the opinion of the site investigator is likely to interfere with evaluation of disease assessment.

  --NOTE: Continuation of hormonal therapies is allowed.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Major surgery ≤ 4 weeks from registration. NOTE: Diagnostic laparoscopy (without other intervention) and/or biopsies (needle aspirate, core biopsy, open biopsy, etc…) are not considered major surgery. If subject received surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Uncontrolled intercurrent illness which in the opinion of the investigator poses unacceptably high risk when combined with study treatment, including but not limited to the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Severely impaired lung function
  * Known history of active TB (Bacillus Tuberculosis)
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN

    ---(NOTE: Optimal glycemic control should be achieved before starting trial therapy.)
  * Significant underlying liver disease such as cirrhosis or severe hepatic impairment
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* For patients in whom planned RT fields will include the heart, any of the following heart conditions, if in the opinion of the investigator they pose unacceptably high risk when combined with study treatment:

  * Prior symptomatic congestive heart failure
  * Documented myocardial infarction ≤6 months prior to registration (pretreatment ECG evidence of infarct only will not exclude patients)
  * Prior significant ventricular arrhythmia requiring medication
  * Prior 2nd or 3rd degree heart block or other types of clinically significant conduction delay ≤ 6 months prior to registration
  * Clinically significant pericardial disease (including pericardial effusion, pericarditis) or cardiac valvular disease ≤12 months prior to registration NOTE: As part of history and physical, all patients must be assessed for signs or symptoms of cardiac disease, or for prior history of cardiac disease. These conditions include but are not limited to diseases related to cardiac valves, pericardium, myocardium, atrioventricular delays or arrhythmias. It is strongly recommended that signs or symptoms of potentially clinically significant disease be evaluated with comprehensive cardiac echo.
* For patients in whom planned RT fields during the study will include the chest, any of the following, if in the opinion of the site investigator they pose unacceptably high risk when combined with study treatment:

  * Prior fistula within thorax, including bronchoalveolar or esophageal.
  * Respiratory condition that required oxygen supplementation ≤ 3 months prior to registration
  * Clinically significant pulmonary hypertension ≤ 12 months prior to registration
  * Pneumonia requiring treatment ≤ 1 month prior to registration
  * Pulmonary embolism requiring treatment ≤ 6 months prior to registration
  * Pleural effusion requiring drainage ≤ 12 months prior to registration
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Currently uncontrolled hyper/hypothyroidism or hyper/hypocortisolism if in the opinion of the investigator they pose unacceptably high risk when combined with study treatment
* Received live vaccine ≤ 30 days prior to registration. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of organ or stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Yoon, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A : Pembrolizumab + External Beam Radiation Therapy: Pembrolizumab + External Beam Radiation Therapy
  Pembrolizumab: 200mg IV at day -21, then day 1 of each 21-day cycle for a maximum of 24 continuous months of Pembrolizumab (35 cycles) from Cycle 1 Day 1 (C1D1) can be administered.
  External Beam Radiation Therapy: 20-30 Gy over five fractions for up to two cycles.
Period: Study Treatment - Up to 22 Months
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Started | 14
Completed | 0
Not Completed | 14
Not completed — Disease Progression | 6
Not completed — Alternative Cancer Therapy | 2
Not completed — AE / Side Effects / Complications | 3
Not completed — Death | 2
Not completed — Symptomatic Deterioration | 1
Period: Follow up - Up to 2 Years
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Started (Treatment and Follow-up are sequential time periods. All subjects from the Treatment time period continue to the follow-up time period, regardless of their completion status.) | 14
Completed | 0
Not Completed | 14
Not completed — Death | 9
Not completed — Patient lost to follow up | 1
Not completed — Patient Refused to follow up | 1
Not completed — study terminated | 1
Not completed — Patient would like to seek treatments locally. | 1
Not completed — Patient stopped protocol treatment due to lack of response to treatment regimen. | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A : Pembrolizumab + External Beam Radiation Therapy: Pembrolizumab + External Beam Radiation Therapy
  Pembrolizumab: 200mg IV at day -21, then day 1 of each 21-day cycle for a maximum of 24 continuous months of Pembrolizumab (35 cycles) from C1D1 can be administered.
  External Beam Radiation Therapy: 20-30 Gy over five fractions for up to two cycles.
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 55.0 [43.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 6
  Carcinoma, NOS | 4
  Squamous Carcinoma | 4
Bone involvement [Count of Participants; unit: Participants]
  Yes | 5
  No | 9
Thoracic involvement [Count of Participants; unit: Participants]
  Yes | 9
  No | 5
Abdominal/Pelvic involvement [Count of Participants; unit: Participants]
  Yes | 13
  No | 1
Total number of metastatic sites [Median (Full Range); unit: number of sites] | 3 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Abscopal Response Rate
Description: Evaluate the abscopal response rate in Carcinoma of Unknown Primary (CUP) patients treated with the combination of pembrolizumab plus radiotherapy. Best abscopal response is defined as the frequency of patients whose best responding abscopal lesion demonstrates at least a 30% decrease in its longest diameter from baseline (Golden et al., 2015).
Time Frame: From Cycle 3, Day 1 (each cycle is 21 days) (C3D1) until death or up to a maximum of 19 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
percentage of participants | 7.1 [0.2 to 33.9]

2. Secondary Outcome: Response Rate
Description: To determine the response rate by RECIST 1.1 and informed by irRECIST, of non-irradiated metastatic sites when pembrolizumab is combined with radiotherapy. Subjects with confirmed CR or PR per RECIST 1.1 should be considered.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until death or up to a maximum of 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Evaluate Treatment-related Toxicity.
Description: The maximum grade for each type of adverse event will be summarized using CTCAE version 4.0 criteria. The frequency and percentage of grade 2+ adverse events will be summarized using CTCAE version 4.0 criteria.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until death or up to a maximum of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
Participants
  Number of patients had at least one adverse event of any grade | 14
  Number of patients had at least one grade 3 or greater adverse event | 8
  Number of patients had at least one grade 3 or greater treatment related adverse event | 5
  Number of patients having serious adverse event | 7

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from registration to the first of either disease progression or death from any cause, where disease progression will be determined based on RECIST 1.1 criteria. Patients that are alive and progression-free will be censored on their last tumor evaluation date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until progression or death or up to a maximum of 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
months | 2.2 [2.0 to NA] — upper limit was not reached due to insufficient number of participants with events.

5. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from registration to death from any cause. Subjects who did not die will be censored at their last visit.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until death or up to a maximum of 19 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
months | 8.2 [2.4 to NA] — upper limit was not reached due to insufficient number of participants with events.

6. Secondary Outcome: Time-to-Progression
Description: Time-to-Progression (TTP) is defined as the time from registration to disease progression, where patients that are progression-free will be censored on their last tumor evaluation date.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until death or up to a maximum of 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
months | 3.5 [2.0 to NA] — upper limit was not reached due to insufficient number of participants with events.

7. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate (DCR) is defined as the frequency (%) of patients who have a best response of PR, CR, or Stable disease based on RECIST 1.1 criteria.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; stable disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum of the longest diameter since the treatment started.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) to a maximum of 19 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 14
percentage of participants | 35.7 [12.8 to 64.9]

8. Secondary Outcome: Explore the Association Between Response Rate (RR) and Other Endpoints (e.g., OS, PFS)
Description: The association between RR (using RECIST 1.1 (informed by irRECIST)) with other clinical endpoints (e.g., OS, PFS, etc.) was performed.
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) until death or up to a maximum of 19 months
Population: Per RECIST 1.1 criteria, no confirmed CR or PR responses were observed.
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Cycle 1, Day 1 (each cycle is 21 days) visit up to a maximum of 19 months.
Description: Adverse events were collected for every subject at every cycle of treatment at an interval of 21 days from the time of consent until 30 days after last dose of Pembrolizumab.
  Serious AE (SAE) at any visit will continue to be followed until the AE resolves to ≤ Grade 1 or baseline, deemed clinically insignificant, and/or until a new anti-cancer treatment starts, whichever is earlier.
Arm/Group | Arm A : Pembrolizumab + External Beam Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A : Pembrolizumab + External Beam Radiation Therapy (N=14)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (3)
SEPSIS (Infections and infestations) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
VASCULAR DISORDERS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A : Pembrolizumab + External Beam Radiation Therapy (N=14)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (5)
ANEMIA (Blood and lymphatic system disorders) | 6 (9)
ANOREXIA (Metabolism and nutrition disorders) | 4 (5)
ANXIETY (Psychiatric disorders) | 3 (4)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
BLOATING (Gastrointestinal disorders) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 2 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE INCREASED (Investigations) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EDEMA LIMBS (General disorders) | 1 (1)
FATIGUE (General disorders) | 4 (5)
FEVER (General disorders) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (4)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPONATREMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOTHYROIDISM (Endocrine disorders) | 3 (4)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INVESTIGATIONS (Investigations) | 2 (8)
LYMPHOCYTE COUNT DECREASED (Investigations) | 6 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (6)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (2)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 1 (2)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (2)
WEIGHT GAIN (Investigations) | 1 (1)
WEIGHT LOSS (Investigations) | 5 (7)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT03396471/Prot_SAP_000.pdf